CLINICAL TRIAL: NCT01253421
Title: The Effects of Dopamine on Reward Processing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Diego A. Pizzagalli, Director, Center for Depression, Anxiety and Stress Research, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-P001568; R01MH068376 (NIH)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: MDD; Major Depressive Disorder; Amisulpride
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Amisulpride

STUDY DESIGN:
Intervention Model Description: There were two groups of subjects: currently experiencing a major depressive episode, or normal health controls. The groups were matched for age, gender, and race. Within each group, half of the subjects were assigned to receive the study drug (amisulpride) and half to receive a placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MDD-amisulpride (Active Comparator): Subjects experiencing a current episode of major depression who are randomized to receive amisulpride
  Interventions: Drug: amisulpride
- MDD-placebo (Placebo Comparator): Subjects experiencing a current episode of major depression who are randomized to receive placebo
  Interventions: Drug: placebo
- HC-amisulpride (Active Comparator): Subjects having no history of mental disorder (healthy controls, HC) who are randomized to receive amisulpride
  Interventions: Drug: amisulpride
- HC-placebo (Placebo Comparator): Subjects having no history of mental disorder who are randomized to receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: amisulpride — single low-dose pharmacological challenge, 50 mg amisulpride
  Other Names: Solian
  Arms: HC-amisulpride; MDD-amisulpride
Drug: placebo — single-dose placebo capsule
  Arms: HC-placebo; MDD-placebo

SUMMARY:
The purpose of this study is to evaluate the effects of a single low dose of the D2/D3 antagonist amisulpride on reward processing. More generally, this study will test the role of dopamine (a naturally occurring brain chemical) in depression.

Hypotheses:

Administration of a single low dose of the D2/D3 antagonist amisulpride will (1) improve performance in a behavioral task assessing learning from feedback and (2) boost activation in reward-related brain regions.

DETAILED DESCRIPTION:
Through an integration of a functional magnetic resonance imaging (fMRI) approach coupled with a pharmacological challenge, the goal of the current study will be to investigate the role of dopamine in MDD. Participants in this research will include 36 MDD subjects and 36 demographically matched healthy participants recruited from the community by Dr. Pizzagalli's laboratory at McLean Hospital's Center for Depression, Anxiety and Stress Research. This study will include two sessions:

* The first session will involve a diagnostic interview, and a series of questionnaires and assessments.
* The second session will take place at the McLean Hospital's Neuroimaging Center, and include the administration of a low-dose of amisulpride (50 mg capsule) or placebo, followed by an fMRI brain scan and administration of two behavioral tasks.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for subjects with Major Depressive Disorder (MDD):

  1. Diagnostic and Statistical Manual of Mental Disorders (DSM IV) diagnostic criteria for MDD, diagnosed with the use of the Structured Clinical Interview for DSM Disorders (SCID);
  2. Written informed consent;
  3. Both genders and all ethnic origins, age between 18 and 45;
  4. A baseline score > 16 on the Hamilton Rating Scale for Depression (HRSD) 17-item version;
  5. Right-handed.
  6. Absence of any psychotropic medications for at least 2 weeks:

     * 6 weeks for fluoxetine,
     * 6 months for neuroleptics,
     * 2 weeks for benzodiazepines,
     * 2 weeks for any other antidepressants.

Inclusion Criteria for Control Subjects:

1. Absence of medical, neurological, and psychiatric illness (including alcohol and substance abuse), as assessed by subject history and a structured clinical interview (SCID-I/NP);
2. Written informed consent;
3. Both genders and all ethnic origins, age between 18 and 45;
4. Right-handed;
5. Absence of any medications for at least 3 weeks;
6. Absence of pregnancy.

Exclusion Criteria:

* Exclusion Criteria for All Subjects:

  1. Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment;
  2. Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, intrauterine device, s/p tubal ligation, or partner with vasectomy);
  3. Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurological or hematologic disease;
  4. Lifetime history of seizure disorder;
  5. Lifetime history or current diagnosis of any of the following DSM-IV psychiatric illnesses: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, substance dependence, substance abuse within the last 12 months (with the exception of alcohol abuse within the last 12 months, which is permissible for MDD subjects); eating disorders, post-traumatic stress disorder (lifetime PTSD is exclusionary for control subjects, PTSD within the last 24 months is exclusionary for MDD subjects); simple phobia, social anxiety disorder and generalized anxiety disorders will be allowed only if secondary to MDD;
  6. More than five instances of lifetime cocaine or stimulant use (e.g., amphetamine, cocaine, methamphetamine);
  7. Use of dopaminergic drugs (including methylphenidate) within the last 6 months;
  8. Lifetime history or current diagnosis of dementia, or a score of < 26 on the Mini Mental Status Examination at the screening visit;
  9. Lifetime history of adverse drug reactions or allergy to the study drug (amisulpride);
  10. Patients with mood congruent or mood incongruent psychotic features;
  11. Current use of other psychotropic drugs;
  12. Clinical or laboratory evidence of hypothyroidism;
  13. Patients with a lifetime history of electroconvulsive therapy (ECT);
  14. Patients with renal insufficiency;
  15. Failure to meet standard MRI safety requirements
  16. Electrolytes, blood urea nitrogen, creatinine: outside the normal range (also ruling out renal insufficiency);
  17. Liver function tests above 1.5 times the upper normal;
  18. Corrected QT interval (QTc) interval in EKG above 450 ms or EKG indicative of arrhythmia or cardiac conduction abnormalities;
  19. Diabetes with poor glucose control;
  20. Cardiac disease, bradycardia less than 55 bpm, hypokalemia, congenital prolongation of QT interval or on-going treatment with a medication likely to induce one of these conditions.
  21. Currently in cognitive-behavioral therapy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Pizzagalli, PhD, Principal Investigator — McLean Hospital, Harvard University
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Admon R, Kaiser RH, Dillon DG, Beltzer M, Goer F, Olson DP, Vitaliano G, Pizzagalli DA. Dopaminergic Enhancement of Striatal Response to Reward in Major Depression. Am J Psychiatry. 2017 Apr 1;174(4):378-386. doi: 10.1176/appi.ajp.2016.16010111. Epub 2016 Oct 24. PMID 27771973
- [Derived] Liu Y, Admon R, Mellem MS, Belleau EL, Kaiser RH, Clegg R, Beltzer M, Goer F, Vitaliano G, Ahammad P, Pizzagalli DA. Machine Learning Identifies Large-Scale Reward-Related Activity Modulated by Dopaminergic Enhancement in Major Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Feb;5(2):163-172. doi: 10.1016/j.bpsc.2019.10.002. Epub 2019 Oct 22. PMID 31784354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at McLean Hospital (Belmont, MA) and Massachusetts General Hospital (MGH; Boston, MA) between February, 2012, and September, 2015. The study was advertised using flyers, and on a number of internet bulletin boards available to the general public. Study visits were conducted in research facilities at McLean Hospital.
Pre-assignment Details: An assessment visit was conducted prior to the drug-challenge visit. Subjects had a diagnostic interview (SCID) and preliminary physical exam, provided a blood sample for lab tests, and completed surveys, to determine eligibility. Those meeting eligibility criteria were scheduled for a drug+scanning visit where randomization occurred.
Groups:
- All Participants Prior to Randomization: All Participants went through Assessment, prior to randomization.
- HC-amisulpride: Subjects having no history of mental disorder who are randomized to receive amisulpride
Period: Assessment and Scheduling
Arm/Group | All Participants Prior to Randomization | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Started (Enrolled for screening visit) | 159 | 0 (Arm has no participants until randomization.) | 0 (Arm has no participants until randomization.) | 0 (Arm has no participants until randomization.) | 0 (Arm has no participants until randomization.)
Eligible After Screening Visit | 85 | 0 | 0 | 0 | 0
Returned for Drug+Scanning Visit (This milestone accounts for participants who were lost to follow up or withdrew for other reasons.) | 60 | 0 | 0 | 0 | 0
Completed (These 60 participants enter Period 2.) | 60 | 0 | 0 | 0 | 0
Not Completed | 99 | 0 | 0 | 0 | 0
Not completed — Found to be Ineligible | 74 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 17 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Period: Drug+Scanning Visit
Arm/Group | All Participants Prior to Randomization | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Started (At the start of this period, all 60 active participants are randomized to a drug-X-condition arm) | 0 (Arm has no participants once randomization has occurred.) | 15 | 14 | 16 | 15
Received Drug Challenge | 0 | 15 | 14 | 16 | 15
Completed | 0 | 15 | 14 | 16 | 14
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- MDD-amisulpride: Subjects experiencing a current episode of major depression who received amisulpride
- MDD-placebo: Subjects experiencing a current episode of major depression who received placebo
- HC-amisulpride: Subjects having no history of mental disorder who received amisulpride
- HC-placebo: Subjects having no history of mental disorder who received placebo
- Total: Total of all reporting groups
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo | Total
Number analyzed (Participants) | 15 | 14 | 16 | 14 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.20 (8.6) | 25.8 (5.35) | 25.3 (25.3) | 24.7 (24.7) | 26 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 11 | 9 | 38
  Male | 3 | 8 | 5 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 3 | 0 | 7
  Not Hispanic or Latino | 12 | 13 | 12 | 14 | 51
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 2 | 2 | 0 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 3 | 9
  White | 11 | 9 | 10 | 6 | 36
  More than one race | 1 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 16 | 14 | 59
Educ-yrs [Mean (Standard Deviation); unit: years] — Years of Education
  years | 15.6 (2.06) | 16.6 (2.90) | 16.2 (2.13) | 16.5 (1.52) | 16.2 (2.18)
Menstrual phase [Count of Participants; unit: Participants] — Menstrual phase when scanned (females only) Population: Percent among females only
  Participants
    number analyzed (Participants) | 12 | 6 | 11 | 9 | 38
    Follicular | 1 | 2 | 6 | 3 | 12
    Luteal | 4 | 1 | 1 | 3 | 9
    Unknown | 7 | 3 | 4 | 3 | 17
HRSD [Mean (Standard Deviation); unit: units on a scale] — Hamilton Rating Scale for Depression (HRSD), 17 item. Range: 0 (no symptoms) to 52 (maximum symptom severity) Clinical categories for total score: 0-7: absent; 8-13: mild; 14-19: moderate; 20-25: severe; 26-52: very severe. Population: 5 missing values
  units on a scale
    number analyzed (Participants) | 14 | 14 | 13 | 13 | 54
    (all) | 16.4 (3.37) | 18.4 (5.09) | 1.0 (1.58) | 0.5 (0.66) | 9.37 (8.997)
MDD SCID rating [Mean (Standard Deviation); unit: units on a scale] — Diagnostic rating of Major Depressive Disorder (MDD): 3=Meets Criteria; 2=Subthreshold; 1=Absent
  units on a scale | 2.9 (.27) | 2.9 (.27) | 1 (0) | 1 (0) | 1.93 (.99)
# MDEs [Mean (Standard Deviation); unit: Episodes] — Number of discrete major depressive episodes (MDE). Population: Applies to MDD subjects only
  Episodes
    number analyzed (Participants) | 15 | 14 | 0 | 0 | 29
    (all) | 2.75 (2.667) | 4.79 (3.490) |  |  | 3.74 (3.230)
Length_MDE [Mean (Standard Deviation); unit: months] — Length of the current major depressive episode (months) Population: Statistics include MDD subjects only
  months
    number analyzed (Participants) | 15 | 14 | 0 | 0 | 29
    (all) | 20.50 (16.53) | 14.00 (18.982) |  |  | 16.17 (17.771)
Patients with comorbid anxiety disorder [Count of Participants; unit: Participants] — Number of subjects with current comorbid Anxiety Disorders
  Participants
    Has comorbid Anxiety Disorder | 3 | 6 | 0 | 0 | 9
    No comorbid Anxiety Disorder | 9 | 8 | 16 | 14 | 47
    Unknown | 3 | 0 | 0 | 0 | 3
Patients with past anxiety disorder [Count of Participants; unit: Participants] — Number of subjects with past comorbid Anxiety Disorders
  Participants
    Yes | 3 | 6 | 0 | 0 | 9
    No | 9 | 8 | 16 | 14 | 47
    Unknown | 3 | 0 | 0 | 0 | 3
TCI Total [Mean (Standard Deviation); unit: units on a scale] — Total score on the Novelty-Seeking (NS) subset of the Temperament and Character Inventory (TCI). The NS subset consists of 35 items from the full 240-item TCI survey.
  ITEMS: statements people might use to describe their attitudes, opinions, interests, and other personal feelings. Item responses are on a 5-point scale of 1 (definitely false) to 5 (definitely true); Range: 35-175.
  Higher scores indicate higher Novelty-Seeking temperament.
  units on a scale | 87.97 (13.992) | 94.2 (17.78) | 103.9 (13.99) | 105.9 (14.53) | 97.97 (16.417)
TCI NS-1 [Mean (Standard Deviation); unit: units on a scale] — TCI NS subscale 1 - "Exploratory excitability v stoic rigidity"; 10 items, Range: 10-50; Higher scores indicate higher degree of exploratory excitability
  units on a scale | 27.760 (5.4779) | 29.385 (5.3000) | 34.200 (5.7595) | 35.857 (5.8159) | 31.814 (6.4070)
TCI NS-2 [Mean (Standard Deviation); unit: units on a scale] — TCI NS subscale 2 - "Impulsiveness v reflection"; 9 items, Range: 9-45; Higher scores indicate higher degree of impulsiveness
  units on a scale | 19.60 (4.137) | 20.85 (6.053) | 22.93 (4.698) | 22.79 (5.860) | 21.54 (5.258)
TCI NS-3 [Mean (Standard Deviation); unit: units on a scale] — TCI NS subscale 3 - "Extravagance v reserve" ; 9 items, Range: 9-45; Higher scores indicate higher degree of extravagance.
  units on a scale | 23.873 (6.9297) | 25.231 (8.8615) | 26.667 (5.5891) | 26.571 (4.3273) | 25.581 (6.5084)
TCI NS-4 [Mean (Standard Deviation); unit: units on a scale] — TCI NS subscale 4 - "Disorderliness v regimentation" ; 7 items, Range: 7-35; Higher scores indicate higher degree of disorderliness.
  units on a scale | 16.73 (3.973) | 18.77 (3.468) | 20.07 (5.311) | 20.64 (4.551) | 19.04 (4.555)
BIS attention-1 [Mean (Standard Deviation); unit: units on a scale] — Attention subscale (first order) of the Barratt Impulsiveness Scale (BIS); 5 items, item responses are on a scale from 1 (not impulsive) to 4 (very impulsive); Range 5-20, higher scores indicate less stable attention
  units on a scale | 10.393 (2.3053) | 9.929 (1.9400) | 9.620 (1.9879) | 11.000 (2.3205) | 10.225 (2.1500)
BIS cognitive instability [Mean (Standard Deviation); unit: units on a scale] — Cognitive Instability subscale (first order) of the BIS; 3 items, item responses are on a scale from 1 (not impulsive) to 4 (very impulsive); Range 3-12, higher scores indicate less stable cognition
  units on a scale | 5.143 (1.7913) | 5.536 (1.9852) | 4.467 (1.1255) | 5.857 (1.5619) | 5.237 (1.6800)
BIS motor-1 [Mean (Standard Deviation); unit: units on a scale] — Motor subscale (first order) of the BIS; 7 items, item responses are on a scale from 1 (not impulsive) to 4 (very impulsive); Range 7-28, higher scores indicate greater motor impulsivity
  units on a scale | 12.714 (2.6144) | 12.786 (2.9136) | 12.133 (2.2636) | 12.071 (2.9733) | 12.421 (2.6454)
BIS perseverance [Mean (Standard Deviation); unit: units on a scale] — Perseverance subscale (first order) of the BIS; 4 items, item responses are on a scale from 1 (not impulsive) to 4 (very impulsive); Range 4-16, higher scores indicate more perseveration
  units on a scale | 6.643 (1.5984) | 6.857 (1.6104) | 6.847 (1.4426) | 7.693 (1.9408) | 7.007 (1.6593)
BIS self control [Mean (Standard Deviation); unit: units on a scale] — Self-control subscale (first order) of the BIS; 6 items, item responses are on a scale from 1 (not impulsive) to 4 (very impulsive); Range 6-24, higher scores indicate less self-control
  units on a scale | 11.071 (3.2455) | 10.429 (3.0813) | 11.067 (3.6345) | 12.357 (3.2959) | 11.228 (3.3113)
BIS cognitive complexity [Mean (Standard Deviation); unit: units on a scale] — Cognitive Complexity subscale (first order) of the BIS; 5 items, item responses are on a scale from 1 (not impulsive) to 4 (very impulsive); range 5-20, higher scores indicate greater difficulty with complexity
  units on a scale | 9.786 (2.0069) | 10.161 (2.9509) | 9.933 (2.3442) | 10.554 (2.4143) | 10.105 (2.4016)
BIS Attention-2 [Mean (Standard Deviation); unit: units on a scale] — Attentional Impulsivity subscale (second order) of the BIS; Sum of the Attention-1 and Cognitive Instability subscales; Range 8-32, higher scores indicate less ability to control attention
  units on a scale | 15.536 (3.6187) | 15.464 (2.7767) | 14.087 (2.8332) | 16.857 (3.2548) | 15.461 (3.2078)
BIS Motor-2 [Mean (Standard Deviation); unit: units on a scale] — Motor impulsivity subscale (second order) of the BIS; Sum of the Motor-1 and Perseverance subscales; Range 11-44, higher scores indicate more impulsive movement
  units on a scale | 19.357 (3.2959) | 19.643 (3.5865) | 18.980 (2.8016) | 19.764 (3.7056) | 19.428 (3.2791)
BIS Non-planning-2 [Mean (Standard Deviation); unit: units on a scale] — Non-planning subscale (second order) of the BIS; Sum of the Self-control and Cognitive Complexity subscales; Range 11-44, higher scores indicate less ability to guide according to a plan
  units on a scale | 20.857 (4.1668) | 20.589 (5.2638) | 21.000 (5.7446) | 22.911 (4.1459) | 21.333 (4.8528)
MASQ total [Mean (Standard Deviation); unit: units on a scale] — Mood and Anxiety Symptom Questionnaire (MASQ), short form. Measures the severity of anxiety and depressive symptoms.
  62 items, rating of how much you have experienced certain feelings, emotions, or behaviors in the past week; item responses are on a 5-point scale from 1 (not at all) to 5 (extremely).
  Range: 62-310; higher scores indicates more severe symptoms.
  units on a scale | 173.727 (14.2367) | 174.077 (18.5448) | 92.350 (16.0618) | 88.571 (12.4389) | 131.476 (44.6597)
MASQ GDA [Mean (Standard Deviation); unit: units on a scale] — General Distress-Anxiety (GDA) subscale of the MASQ. 11 items on a scale of 1 to 5. Range: 11-55, higher scores indicate greater severity of anxiety symptoms.
  units on a scale | 21.800 (6.2244) | 23.385 (6.7520) | 14.200 (3.3209) | 12.071 (1.9793) | 17.772 (6.8060)
MASQ GDD [Mean (Standard Deviation); unit: units on a scale] — General Distress-Depression (GDD) subscale of the MASQ. 12 items on a scale of 1 to 5. Range: 12-60, higher scores indicate greater severity of depressive symptoms.
  units on a scale | 41.960 (7.7346) | 39.538 (7.2872) | 14.533 (3.6029) | 14.214 (2.9136) | 27.375 (14.5034)
MASQ AA [Mean (Standard Deviation); unit: units on a scale] — Anxious Arousal (AA) subscale of the MASQ; 17 items on a scale of 1 to 5; Range: 17-85, higher scores indicate greater severity of anxious arousal symptoms.
  units on a scale | 21.880 (2.9644) | 23.385 (4.4260) | 19.417 (3.3643) | 17.643 (1.1507) | 20.534 (3.7852)
MASQ AD [Mean (Standard Deviation); unit: units on a scale] — Anhedonic Depression (AD) subscale of the MASQ; 22 items on a scale of 1 to 5; Range: 22-110, higher scores indicate greater severity of anhedonic symptoms.
  units on a scale | 88.087 (9.1143) | 87.769 (6.9180) | 44.200 (8.4448) | 44.643 (9.6764) | 65.795 (23.5064)
RSES_Total [Mean (Standard Deviation); unit: units on a scale] — Rosenberg Self Esteem Scale (RSES) total score. A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. All items are answered using a Likert scale ranging from strongly disagree (0) to strongly agree (3); scores on negative feelings are inverted.
  Range: 0-30, higher scores indicate higher self-esteem.
  units on a scale | 26.36 (4.802) | 26.36 (5.988) | 14.14 (3.891) | 14.33 (4.633) | 21.86 (7.651)
Defeat Scale [Mean (Standard Deviation); unit: units on a scale] — The level of defeat-related feelings the participant has felt in the past week. 16 items, rated on a scale from 0 (never) to 4 (always). Range: 0 to 64; higher scores indicate greater feelings of defeat.
  units on a scale | 38.09 (6.700) | 35.55 (9.720) | 5.88 (3.182) | 5.25 (5.392) | 23.66 (17.049)
BDI-II [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory-II (BDI-II). Measures the presence and severity of 21 depressive symptoms during the past two weeks, on a scale from 0 (none, or no change) to 3 (persistent, or worsening).
  Range: 0 to 63. Higher scores indicate greater symptom severity. Clinical categories for total score: 0-14: absent; 14-19: mild; 20-28: moderate; 29-63: severe.
  units on a scale | 24.40 (8.423) | 27.91 (7.877) | 1.31 (2.387) | 1.51 (3.131) | 13.54 (13.828)
SHPS total [Mean (Standard Deviation); unit: units on a scale] — Snaith Hamilton Pleasure Scale (SHPS); assesses capacity to experience pleasure (hedonic tone).
  Items: 35 statements that a person might enjoy a particular activity. Item responses are on a 4-point scale of 1 (Strongly agree) to 4 (Strongly disagree).
  Range: 35-140, higher scores indicate greater anhedonia.
  units on a scale | 32.753 (4.6489) | 32.450 (7.5103) | 21.293 (5.6623) | 23.714 (7.4258) | 27.534 (8.0970)
SHPS-low [Mean (Standard Deviation); unit: Count of 'low' responses (1 or 2)] — Number of "low" responses (value is 1 or 2) on the SHPS. Range: 0-14; higher scores indicate better hedonic tone.
  Count of 'low' responses (1 or 2) | 7.667 (1.3452) | 6.857 (1.0995) | 6.400 (1.8439) | 6.571 (2.9013) | 6.879 (1.9293)
AES [Mean (Standard Deviation); unit: units on a scale] — Apathy Evaluation Scale (AES), assesses apathy during the past 4 weeks. Items: 18 statements about a person feeling interest, initiative, or motivation. Item responses are on a 4-point scale of 1 (Not at all true) to 4 (Very true).
  Range: 18-72, lower scores indicate greater apathy.
  units on a scale | 43.45 (7.063) | 42.14 (4.786) | 59.53 (4.856) | 60.86 (4.400) | 51.63 (10.218)
Current smokers [Count of Participants; unit: Participants] — Number of current smokers per group
  Participants | 0 | 0 | 0 | 0 | 0
Past smokers [Count of Participants; unit: Participants] — Number of subject who were smokers in the past
  Participants | 0 | 1 | 0 | 0 | 1
Current drinkers [Count of Participants; unit: Participants] — Number of subjects who drink alcoholic beverages
  Participants | 4 | 6 | 5 | 4 | 19
Drinks in past 24hrs [Mean (Standard Deviation); unit: equivalent shot/can/glasses] — Average number of drinks in the past 24 hours
  equivalent shot/can/glasses | 0.29 (0.469) | 0.46 (0.519) | 0.36 (0.497) | 0.29 (0.469) | 0.35 (0.480)
Usual caffeine (mg) [Mean (Standard Deviation); unit: milligrams] — Amount of caffeine consumed on a normal day in milligrams
  milligrams | 124.35 (74.162) | 176.50 (87.444) | 82.93 (77.308) | 64.75 (41.139) | 111.05 (111.05)
Caffeine today (mg) [Mean (Standard Deviation); unit: milligrams] — Amount of caffeine consumed on the day of testing in milligrams
  milligrams | 81.23 (83.400) | 102.88 (108.938) | 32.13 (32.335) | 67.23 (67.268) | 69.44 (79.159)

OUTCOME MEASURES:

1. Primary Outcome: Effect on PST Reward Learning
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on the ability to learn from rewards during a Probabilistic Selection Task (PST). A higher effect size indicates greater ability to learn from reward trials.
Time Frame: administered after scan
Population: Reward-learning results are missing for 7 subjects
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 14 | 12 | 15 | 11
Effect size (Beta) | 0.6271 (0.15608) | 0.7575 (0.1676) | 0.823 (0.1228) | 0.7545 (0.1828)

2. Primary Outcome: Effect on PST Penalty Learning
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on the ability to learn from penalties during a Probabilistic Selection Task (PST). A higher effect size indicates greater ability to learn from penalty trials.
Time Frame: administered after scan
Population: Penalty-learning results are missing for 7 subjects
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 14 | 12 | 15 | 11
Effect size (Beta) | 0.2428 (0.1800) | 0.29 (0.2056) | 0.2207 (0.20225) | 0.2391 (0.14618)

3. Primary Outcome: Effect on Caudate Response to Cues
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on caudate activation after presentation of a cue. Positive values indicate an increase in activation relative to baseline.
Time Frame: Scan session
Population: Data are missing for 8 subjects due to poor MRI quality.
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 13 | 11 | 16 | 11
Effect size (Beta) | 0.2231 (0.42189) | -0.0391 (0.32792) | -0.0938 (0.57788) | 0.0582 (0.30318)

4. Primary Outcome: Effect on NAcc Response to Cues
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on nucleus accumbens (NAcc) activation after presentation of a cue. Positive values indicate an increase in activation relative to baseline.
Time Frame: Scan session
Population: Data are missing for 8 subjects due to poor MRI quality
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 13 | 11 | 16 | 11
Effect size (Beta) | 0.2446 (0.38546) | 0.0736 (0.38694) | 0.1356 (0.51800) | 0.2182 (0.55236)

5. Primary Outcome: Putamen Response to Cues
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on putamen activation after presentation of a cue. Positive values indicate an increase in activation relative to baseline.
Time Frame: Scan session
Population: Data are missing for 9 subjects due to poor MRI quality
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 13 | 11 | 16 | 10
Effect size (Beta) | 0.4969 (0.41086) | 0.3955 (0.36653) | 0.4169 (0.41839) | 0.3808 (0.42303)

6. Primary Outcome: Effect on Caudate Response to Reward
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on caudate activation after Reward outcomes. Positive values indicate an increase in activation relative to baseline.
Time Frame: During scan session
Population: Data are missing for 9 subjects due to poor MRI quality
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 12 | 11 | 16 | 11
Effect size (Beta) | 0.5783 (1.0104) | -0.2673 (0.1575) | -0.33 (1.243) | 0.1955 (0.1101)

7. Primary Outcome: Effect on NAcc Response to Reward
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on nucleus accumbens (NAcc) activation after reward outcomes. Positive values indicate an increase in activation relative to baseline.
Time Frame: During scan session
Population: Data are missing for 10 subjects due to poor MRI quality
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 13 | 10 | 16 | 10
Effect size (Beta) | 0.9377 (0.1357) | 0.1578 (0.8534) | 0.4018 (1.2619) | 0.954 (1.0833)

8. Primary Outcome: Effect on Putamen Response to Reward
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on putamen activation (beta) after reward outcomes. Positive values indicate an increase in activation relative to baseline.
Time Frame: During scan session
Population: Data are missing for 9 subjects due to poor MRI quality
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 13 | 11 | 16 | 10
Effect size (Beta) | 0.6338 (0.8394) | 0.1709 (0.7996) | -0.14 (1.2282) | 0.436 (0.6689)

9. Secondary Outcome: Effect on Caudate-dACC Connectivity After Reward
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on functional connectivity between caudate and dorsal anterior cingulate cortex (dACC) in response to reward outcomes
Time Frame: During scan session
Population: Data missing for 8 subjects due to poor MRI quality
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 14 | 11 | 13 | 13
Effect size (Beta) | 0.3628 (0.4057) | 0.3881 (0.3415) | 0.2992 (0.49098) | 0.6192 (0.4270)

10. Secondary Outcome: Effect on NAcc-MCC Connectivity After Reward
Description: This statistic shows the effect (beta) that the combination of diagnosis and drug has on functional connectivity between nucleus accumbens (NAcc) and mid-cingulate cortex (MCC) in response to reward outcomes.
Time Frame: During scan session
Population: Data missing for 8 subjects due to poor MRI quality
Measure: Mean (Standard Deviation); unit: Effect size (Beta)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
Number analyzed (Participants) | 14 | 11 | 13 | 13
Effect size (Beta) | 0.4375 (0.4163) | 0.324 (0.4992) | 0.4846 (0.6279) | 0.4877 (0.5070)

ADVERSE EVENTS:
Time Frame: Full study duration (2012-2015)
Arm/Group | MDD-amisulpride | MDD-placebo | HC-amisulpride | HC-placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/16 | 0/14

LIMITATIONS AND CAVEATS:
The choice of a 50-mg dose of amisulpride was based on animal work showing low doses potentiate striatal dopamine release, have strong hedonic effects, and increase the incentive value of environmental cues. Higher doses may have different results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No